CLINICAL TRIAL: NCT02186288
Title: Effect of High-flow Nasal Cannula Oxygen on Lung Volumes Determined by Electrical Impedance Tomography
Acronym: OXIDIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0196
Record Dates: First submitted 2014-06-20; First posted 2014-07-10 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Critical Care; High-flow Nasal Cannula Oxygen; Electrical Impedance Tomography; End Expiratory Lung Volume; End Expiratory Lung Impedance; Diaphragmatic Ultrasound
Keywords: Critical Care; High-flow nasal cannula oxygen; Electrical impedance tomography; End expiratory lung volume; End expiratory lung impedance; Diaphragmatic ultrasound

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Adult ICU patients
  Interventions: Other: High-flow nasal cannula oxygen

INTERVENTIONS:
Other: High-flow nasal cannula oxygen

SUMMARY:
Effect of High-flow nasal cannula oxygen on end-expiratory lung volumes determined by electrical impedance tomography

DETAILED DESCRIPTION:
Prospective clinical study in ICU with patients requiring High-flow nasal cannula oxygen comparing lung volumes determined by electrical impedance tomography and diaphragmatic ultrasound before, during and after High-flow nasal cannula oxygen.

Duration of High-flow nasal cannula oxygen is 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* • Adult ICU patients requiring High-flow nasal cannula oxygen

  * Consent of patients or family
  * Arterial line

Exclusion Criteria:

* • Tracheotomized patients

  * Dressings in the thoracic area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
End-expiratory lung volume (EELV) determined by electrical impedance tomography before NIV non invasive ventilation | at day 1
End-expiratory lung volume (EELV) determined by electrical impedance tomography during NIV non invasive ventilation | at day 1
End-expiratory lung volume (EELV) determined by electrical impedance tomography after NIV non invasive ventilation | at day 1

SECONDARY OUTCOMES:
Anterior, medio-anterior, medio-posterior and posterior EELV at each time | at day 1
Diaphragmatic excursion and thickness determined by ultrasound | at day 1
Ventilatory frequency | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France